CLINICAL TRIAL: NCT02655861
Title: Prospective Evaluation of Infants and Children With Congenital Ichthyosis
Brief Title: A Multi-center, Prospective Evaluation of Infants and Children With Congenital Ichthyosis
Status: Terminated | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Foundation for Ichthyosis & Related Skin Types (FIRST) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1504015620
Record Dates: First submitted 2015-11-16; First posted 2016-01-14 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Ichthyosis
MeSH Terms: conditions — Ichthyosis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva or blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ichthyosis
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
This project will follow babies with ichthyosis over time in order to better understand the natural course of ichthyosis in infants and children and to examine how specific genetic mutations affect clinical characteristics.

DETAILED DESCRIPTION:
The investigators hypothesize that early complications and comorbidities in infants with congenital ichthyosis are genotype-dependent, such that clinical standards of care can be tailored to the genetic diagnoses. Definition of clinical groups based upon phenotype may also provide useful predictors of outcome. Information gained from this study will provide the basis for the development of rational standards of care for the future management of children with congenital ichthyosis.

ELIGIBILITY:
Inclusion Criteria:

* One parent must be able to understand and sign an informed consent document.
* Newborns who present at or within 2 months of birth with a clinical diagnosis of ichthyosis.
* Families must consent to providing DNA for genetic analysis
* Families must agree to the intake evaluation followed by 10 follow-up evaluations, which will occur at ages 1, 2, 3, 6, 9, 12, 18, 24, and 36 months.

Exclusion Criteria:

* Subjects with non-English speaking parents
* Patients with a family history of ichthyosis vulgaris
* Patients with X-linked ichthyosis

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns who present at or within 2 months of birth with a clinical diagnosis of ichthyosis, except for infants with a family history of ichthyosis vulgaris and infants with X-linked ichthyosis.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-06; Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Weight | 36 Months
  To assess growth, birth weight and all weights (in pounds) obtained during hospitalization and clinic visits will be recorded. The primary outcome of the study will be to determine incidence, timing and severity of "growth failure" in neonates with ichthyosis in relation to genotype at the 3 year pediatric visit. Weight of the child will primarily be used to make this determination.
Length (Height) | 36 Months
  To assess growth, birth length and all subsequent measures (in inches) obtained during hospitalization and clinic visits will be recorded. The primary outcome of the study will be to determine incidence, timing and severity of "growth failure" in neonates with ichthyosis in relation to genotype at the 3 year pediatric visit. Length of the child will primarily be used to make this determination.

SECONDARY OUTCOMES:
Weight | Birth (baseline), 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months
  To assess growth, birth weight and all weights (in pounds) obtained during hospitalization and clinic visits will be recorded. Weight of the child will be used to characterize growth over the course of the 3 year follow up time.
Length (Height) | Birth (baseline), 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months
  To assess growth, birth length and all subsequent measures (in inches) obtained during hospitalization and clinic visits will be recorded. Length of the child will be used to characterize growth over the course of the 3 year follow up time.
Electrolyte Disturbance | Birth (baseline), 1 month, 2 months, 3 months, 12 months, 24 months, 36 months
  Measurements of electrolytes, including calcium, phosphate, magnesium, BUN and creatinine values will be used to evaluate the incidence, timing, and severity of electrolyte disturbances and the management of these disturbances in the neonatal period in relation to phenotypic group and to genotype. This outcome will be captured as a 'yes/no' for any or all of the above.
Systemic Infections | Birth (baseline), 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months
  The incidence, severity timing, and causative organisms of systemic infections during neonatal hospital stays will be reviewed in relation to management, including skin care practices and nursing procedures (e.g., open bed vs. humidified isolette).
Complications of Congenital Ichthyosis | Birth (baseline), 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months
  Clinical severity will be rated using a standardized instrument. The evolution of skin phenotype will be documented via serial standardized photography. Transepidermal Water Loss (TEWL) will be measured in some sites.
Developmental Delays | Birth (baseline), 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months
  To determine the incidence and severity of development delays in relation to genotype, a development history will be obtained at each follow-up evaluation, including information regarding relevant interventions such as physical or occupational therapy. Physical examination at each visit will assess range of motion of digital and major limb joints. This outcome will be captured as a 'yes/no' for any or all of the above.

OTHER OUTCOMES:
Ear and Eye Conditions | Birth (baseline), 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months
  To determine the incidence and severity of ear and eye problems in early childhood in relation to genotype, caregivers will be queried regarding buildup of ear debris and palpebral closure during sleep. Physical exams will assess ear canal patency, lid closure, and signs of conjunctival irritation. If participants are evaluated and/or treated by ophthalmology and otolaryngology, these records will be obtained. This outcome will be captured as a 'yes/no' for any or all of the above.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Criaglow, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States